CLINICAL TRIAL: NCT01195792
Title: A 35-Day, Multi-Centre, Randomised, Parallel-Group, Double-Blind, Placebo-Controlled Proof of Concept Study to Investigate the Effects of GSK1521498 on Body Weight and Composition, Eating Behaviour and Related Brain Function, in Obese Subjects With Over-Eating Behaviours.
Brief Title: A 35 Day Study to Investigate the Effects of GSK1521498 on Bodyweight in Obese Subjects With Over-Eating Behaviours.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111850
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Obesity
Keywords: Opioid receptors; Body weight; Over-eating behaviour; Obesity; Fat mass
MeSH Terms: conditions — Obesity; Body Weight | interventions — N-((3,5-difluoro-3'-(1H-1,2,4-triazol-3-yl)-4-biphenylyl)methyl)-2,3-dihydro-1H-inden-2-amine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2 mg GSK1521498 (Experimental): Approximately 20 subjects will be randomised to receive 2 mg GSK1521498. The drug is being developed for the treatment of obesity due to excessive consumption of high calorie foods
  Interventions: Drug: GSK1521498
- 5 mg GSK1521498 (Experimental): Approximately 20 subjects will be randomised to receive 5 mg GSK1521498. The drug is being developed for the treatment of obesity due to excessive consumption of high calorie foods
  Interventions: Drug: GSK1521498
- Placebo (Placebo Comparator): Approximately 20 subjects will be randomised to receive matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK1521498 — GSK1521498 2mg or 5mg will be given for up to 35 days and subjects will be assessed weekly
  Arms: 2 mg GSK1521498; 5 mg GSK1521498
Drug: Placebo — Placebo will be given for up to 35 days and subjects will be assessed weekly
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether GSK1521498 will cause weight loss in obese but otherwise healthy subjects with over-eating behaviours.

DETAILED DESCRIPTION:
This study is to test a new drug which may be used for treating over-eating behaviours and patterns that some overweight and obese people find difficult to control. The drug works by inhibiting the effects of messenger molecules called opioids. These opioids are naturally produced within the human body, and are involved in controlling how much we eat, and the pleasure we get from eating. We believe that GSK1521498 might be effective in the treatment of obesity because it is well known that drugs working on similar binding sites in the brain reduce the pleasure we get from eating, especially high fat or high sugar food. We also believe the effects of GSK1521498 will be greater in obese individuals with greater severity of over-eating behaviours, as measured for example by existing questionnaire scales for binge-eating or compulsive eating behaviour. We will perform a variety of simple tests using a computer, questionnaires and eating assessments to examine effects on behaviour. We will also ask people to complete questionnaires so that we can see if there are any effects on their mood.

ELIGIBILITY:
Inclusion Criteria:

* Obese but essentially healthy male or female between 18 and 60 years of age inclusive.
* Body Mass Index greater than or equal to 30 kg/m2.
* Binge Eating Scale (BES) score that is greater than or equal to 19 at screening assessment.
* A female subject of child-bearing potential must use one of the contraception methods listed in the protocol prior to the start of the study until at least 14 days after receiving the last dose of study medication.
* Male subjects must agree to use one of the contraception methods listed in the protocol from the time of the first dose of study medication until at least 5 days after receiving the last dose of study medication.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the information sheet or informed consent form. A good understanding of English is required due to the high number of questionnaires and assessments that subjects are required to undergo.
* Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) < 2x Upper limit of Normal (ULN); alkaline phosphatase and bilirubin <1.5x (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Must be right handed (a requirement to ensure consistency of functional magnetic resonance imaging (fMRI) signals from the brain)

Exclusion Criteria:

* Has a history of clinically significant medically diagnosed eating disorders (diagnosed and/or treated) as assessed by Diagnostic and Statistical Manual of Mental Disorders (DSM-IV/V) criteria using the Mini International Neuropsychiatric Interview (MINI).
* Self-administered Beck Depression Inventory II scale total score greater than 13 or suicide question score greater than zero at screening.
* Current history (in the last 6 months) of any Axis 1 psychiatric disorder as assessed by DSM-IV/V criteria using the MINI.
* Subject who, in the investigator/designee's judgement, poses a significant suicide risk. Evidence of serious suicide risk may include any history of suicidal behaviour and/or any evidence of suicidal ideation on any questionnaires e.g. type 4 or 5 on the Columbia Suicide Severity Rating Scale (C-SSRS) in the last 6 months.
* History of substance abuse or dependence in the 6 months prior to screening, as determined by the Investigator/designee or MINI.
* History of regular high level of alcohol consumption.
* Positive pre-study drug/alcohol screen.
* Smoking history that includes regular use of tobacco or nicotine-containing products within 3 months prior to screening
* Use of prohibited medications.
* use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 14 days prior to the first dose of study medication.
* Subjects who do not currently show stable bodyweight, as judged by the PI/designee (e.g. >5% change within the last 3 months)
* Pregnant or lactating females
* Medical history, concurrent medical condition or laboratory result which makes the subject unsuitable for the study. This includes T1 or T2 diabetes mellitus (Fasting Blood Glucose (FBG) >7 mmol/L), untreated dyslipidaemia (fasting lipid profile with a Low Density Lipoprotein (LDL) cholesterol > 5 mmol/L), uncontrolled hypertension
* History of bariatric surgery for obesity.
* QTcB or QTcF > 450 msec.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Current or chronic history of neurological disorders.
* A positive test for HIV or Hepatitis C.
* Sleep apnoea
* Gastrointestinal disease including inflammatory bowel disease, chronic diarrhea, Crohn's or malabsorption syndromes within the past year
* Participated in a clinical trial and has received an investigational product within 90 days.
* Any contraindications or logistical complications anticipated in relation to Magnetic Resonance Imaging (MRI) scanning or other endpoint assessments, including: presence of a cardiac pacemaker or other electronic device or ferromagnetic metal foreign bodies, claustrophobia, inability to lie still on back, waist circumference of more than 170 cm or body weight exceeding maximum capacity of MRI scanners (180 kg).
* Special dietary requirements (e.g. vegetarians, vegans, religious, food-intolerant diets).
* Unsuitable for cannulation.
* Subjects planning to start a calorie controlled diet or major exercise routine.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Clinically and statistically significant weight loss | 35 days

SECONDARY OUTCOMES:
To see if effects on bodyweight are associated with effects on fat mass, eating behaviour brain function and blood and urine markers | 35 days
To see if effects on bodyweight correlate with over-eating behaviour at baseline | 35 days
Safety: adverse events,blood pressure, heart rate, ECG, clinical chemistry, hematology, urinalysis, change in cognition (eg reaction times), change in mood scales, change in neuropsychiatric symptoms | 35 days
Pharmacokinetic/Pharmacodynamic (PK/PD) relationships: effects on primary and secondary outcomes, including estimation of possible dose-response relationships | 35 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United Kingdom (3):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, Birmingham, West Midlands
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Chamberlain SR, Mogg K, Bradley BP, Koch A, Dodds CM, Tao WX, Maltby K, Sarai B, Napolitano A, Richards DB, Bullmore ET, Nathan PJ. Effects of mu opioid receptor antagonism on cognition in obese binge-eating individuals. Psychopharmacology (Berl). 2012 Dec;224(4):501-9. doi: 10.1007/s00213-012-2778-x. Epub 2012 Jul 3. PMID 22752384
- [Background] Ziauddeen H, Chamberlain SR, Nathan PJ, Koch A, Maltby K, Bush M, Tao WX, Napolitano A, Skeggs AL, Brooke AC, Cheke L, Clayton NS, Sadaf Farooqi I, O'Rahilly S, Waterworth D, Song K, Hosking L, Richards DB, Fletcher PC, Bullmore ET. Effects of the mu-opioid receptor antagonist GSK1521498 on hedonic and consummatory eating behaviour: a proof of mechanism study in binge-eating obese subjects. Mol Psychiatry. 2013 Dec;18(12):1287-93. doi: 10.1038/mp.2012.154. Epub 2012 Nov 13. PMID 23147384
- [Derived] Cambridge VC, Ziauddeen H, Nathan PJ, Subramaniam N, Dodds C, Chamberlain SR, Koch A, Maltby K, Skeggs AL, Napolitano A, Farooqi IS, Bullmore ET, Fletcher PC. Neural and behavioral effects of a novel mu opioid receptor antagonist in binge-eating obese people. Biol Psychiatry. 2013 May 1;73(9):887-94. doi: 10.1016/j.biopsych.2012.10.022. Epub 2012 Dec 14. PMID 23245760
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 111850 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111850 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111850 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111850 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111850 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111850 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111850 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register